CLINICAL TRIAL: NCT00002487
Title: INTRAPERITONEAL METHOTREXATE AND DIPYRIDAMOLE AS SALVAGE TREATMENT FOR ADVANCED OVARIAN CARCINOMA
Brief Title: Methotrexate Plus Dipyridamole in Treating Patients With Advanced Ovarian Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ottawa Regional Cancer Centre (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000077374; CAN-OTT-9017; NCI-V92-0012
Record Dates: First submitted 1999-11-01; First posted 2004-08-30 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2000-04

CONDITIONS: Ovarian Cancer
Keywords: recurrent ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Dipyridamole; Methotrexate

INTERVENTIONS:
Drug: dipyridamole
Drug: methotrexate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Dipyridamole may increase the effectiveness of methotrexate and kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining methotrexate and dipyridamole in treating patients with advanced ovarian cancer that is recurrent after or refractory to cisplatin-based chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the clinical complete and partial response rate, pathological complete response rate, disease-free survival, and duration of response produced by intraperitoneal dipyridamole/methotrexate (DP/MTX) administered as a 7-day continuous infusion in patients with advanced ovarian carcinoma that is recurrent following or refractory to cisplatin-based chemotherapy. II. Determine the peritoneal and systemic toxicity of DP/MTX.

OUTLINE: Nonrandomized study. Single-Agent Chemotherapy with Chemopotentiation. Methotrexate, MTX, NSC-740; with Dipyridamole, DP, NSC-515776.

PROJECTED ACCRUAL: Up to 40 evaluable patients in each category (prior intraperitoneal vs. prior intravenous platinum-based chemotherapy) will be studied. If no responses are seen in the first 20 patients in either category, accrual to that category will cease. An accrual rate of 15 patients/year is anticipated.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven, Stage III/IV ovarian carcinoma that is refractory or recurrent within 1 year of complete response to intraperitoneal or intravenous platinum-based chemotherapy Debulking surgery must have been considered at the completion of prior chemotherapy (failure to debulk does not exclude) Clinical or radiographic evidence of advanced, predominantly peritoneal disease on physical exam, CT or MRI scan, exploratory laparotomy, or peritoneal cytology or by elevated CA-125 (above 35 units in Ottawa Civic or General Hospitals) required Disease limited to peritoneal cavity not required, but peritoneal disease should constitute the main life-threatening or symptom-producing component Good distribution of contrast medium throughout peritoneal cavity on CT of abdomen and pelvis required Measurable, evaluable, or unevaluable disease of any size acceptable

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Not specified Life expectancy: More than 2 months Hematopoietic: WBC at least 3,000 Platelets at least 100,000 Hepatic: Bilirubin less than 3 X ULN SGOT less than 3 x ULN Renal: Creatinine less than 1.7 mg/dl (150 micromoles/liter) BUN less than 42 mg/dl (15 mmoles/liter) Other: No requirement for DP or MTX or any medication known to interact with DP, (i.e., antiplatelet or anticoagulant drugs) or MTX (i.e., chemotherapeutic agents) No second malignancy other than basal cell carcinoma of the skin

PRIOR CONCURRENT THERAPY: Recovery from toxicities of prior therapy required Biologic therapy: Not specified Chemotherapy: Prior platinum-based chemotherapy required No concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior abdominopelvic or pelvic radiotherapy No concurrent peritoneal radiotherapy Surgery: See Disease Characteristics Other: No concurrent antiplatelet or vasodilatory agents

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1991-07

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh Goel, MD, FRCPC, Study Chair — Ottawa Regional Cancer Centre
Locations (2):
- Canada (2):
  - Ottawa Regional Cancer Center - General Division, Ottawa, Ontario
  - Ottawa Regional Cancer Centre - Civic Campus, Ottawa, Ontario